CLINICAL TRIAL: NCT00419146
Title: A Multicentre, Placebo-controlled Trial of Eicosapentaenoic Acid (EPA) and Antioxidant Supplementation in the Treatment of Schizophrenia and Related Disorders
Brief Title: Treatment of Schizophrenia With an Omega-3 Fatty Acid (EPA) and Antioxidants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Aker (Other)
Collaborators: Diakonhjemmet Hospital (Other); Stanley Medical Research Institute (Other); Laxdale Ltd (Unknown); Scandinavian Society for Psychopharmacology (Unknown); Shipowner Emil Stray's legacy (Unknown); Johanne and Einar Eilertsen's research fund (Unknown); AstraZeneca (Industry); Solveig and Johan P. Sommer's foundation (Unknown); Josef and Haldis Andresen's legacy (Unknown); University of Oslo (Other); Norwegian University of Science and Technology (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LA.01.07.0001; 01T-106 (Stanley M.R.I.,USA)
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorder; Psychotic Disorders
Keywords: Schizophrenia; Schizophreniform disorders; Schizoaffective disorder; Psychotic disorders; Randomized Controlled Trials; Longitudinal Studies; Fatty Acids, Omega-3; Eicosapentaenoic Acid; Vitamins; Antioxidants; Ascorbic Acid; Alpha-Tocopherol; Placebos; Antipsychotic Agents; Oxidative Stress; Fatty Acids, Unsaturated; Phospholipases; Niacin; Adverse effects; Delusions; Hallucinations; Neuropsychological Tests; Attention; Memory; Hypertriglyceridemia; Models, Statistical
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions; Hallucinations; Hypertriglyceridemia | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ethyl EPA (active) and Vitamins E + C (active) (Experimental)
  Interventions: Drug: Ethyl-eicosapentaenoic acid (EPA); Drug: Vitamins E + C
- Ethyl EPA (active) and Vitamins E+C (placebo) (Experimental)
  Interventions: Drug: Ethyl-eicosapentaenoic acid (EPA); Other: Vitamins E+C (placebo)
- Ethyl EPA (placebo) and Vitamins E+C (active) (Experimental)
  Interventions: Drug: Vitamins E + C; Other: Etyl EPA (placebo)
- Ethyl EPA (placebo) and Vitamins E+C (placebo) (Placebo Comparator)
  Interventions: Other: Vitamins E+C (placebo)

INTERVENTIONS:
Drug: Ethyl-eicosapentaenoic acid (EPA) — Capsules, 2 g per day for 16 weeks
  Other Names: Provided by Laxdale Ltd., Scotland, UK
  Arms: Ethyl EPA (active) and Vitamins E + C (active); Ethyl EPA (active) and Vitamins E+C (placebo)
Drug: Vitamins E + C — RRR-alpha-tocopherol 392 mg + slow-release ascorbic acid 1000 mg per day, for 16 weeks
  Other Names: CellaVie (Ferrosan AS, Denmark)
  Arms: Ethyl EPA (active) and Vitamins E + C (active); Ethyl EPA (placebo) and Vitamins E+C (active)
Other: Etyl EPA (placebo) — Paraffin oil. Capsules, each 0.5 g.
  Other Names: Placebo EPA
  Arms: Ethyl EPA (placebo) and Vitamins E+C (active)
Other: Vitamins E+C (placebo) — Tablets containing dicalciumphosphate
  Other Names: Placebo CellaVie, provided by Ferrosan AS, Denmark
  Arms: Ethyl EPA (active) and Vitamins E+C (placebo); Ethyl EPA (placebo) and Vitamins E+C (placebo)

SUMMARY:
The purpose of this trial is to study the effect of adding the omega-3 fatty acid EPA and/or Vitamins E + C to antipsychotic drugs in younger patients with schizophrenia and related psychoses.

DETAILED DESCRIPTION:
Objective:

Study the effect of adding Ethyl-EPA and/or Vitamins E + C to antipsychotic drugs in younger patients with schizophrenia and related psychoses.

Methods and material:

* Design: Multicentre, randomized, double-blind, placebo-controlled, fixed dose, 2x2 factorial, add-on clinical trial.
* Sample:

  * Patients with schizophrenia, schizoaffective disorder or schizophreniform disorder (DSM-IV); aged 18-40 years; less than 15 years since first psychotic symptoms;admitted to a psychiatric department within the previous 21 days before screening; speaks fluently a Scandinavian language;treated with antipsychotics; written informed consent;no known allergy to trial agents;no substance dependence (DSM-IV);no warfarin currently or anamnestic indicators of impaired haemostasis. Planned: 200 patients. Actually included: 99 intent-to-treat patients.
  * Healthy controls: aged 18-40 years;no mental disorder (DSM-IV). Included: 20 persons.
* Clinical assessments: Positive and Negative Syndrome Scale (PANSS) (main outcome variable). Self-report questionnaire. Adverse effects (UKURS). Neurocognitive assessment battery. Niacin skin flush test. General medical assessment.
* Blood samples: RBC fatty acids, S-α-tocopherol, F2-isoprostane (kits), monocyte mRNA Phospholipase A22 (PLA2) Gr4a and 6a (RT-PCR method), RBC Gr4a PLA2 concentration (ELISA technique), a range of other biochemical tests.
* Experimental treatment over 16 weeks: Ethyl-EPA 2 g/d or Placebo EPA and Vitamin E 364 mg/d + Vitamin C 1000 mg/d or Placebo Antioxidants
* Statistics: Linear Mixed Model for longitudinal analyses of effects; other uni- and multivariate methods (SPSS 12.0 - PASW Statistics 18).

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia, schizophreniform disorder or schizoaffective disorder (DSM-IV)
* Admitted to a psychiatric hospital/department within the previous twenty-one days before screening
* Less than fifteen years, in retrospect, since first psychotic symptoms (DSM-IV 295, criteria A,1-4)
* Age 18-40 years
* Speaks fluently a Scandinavian language
* A written informed consent must be obtained before any trial-related activities

Exclusion Criteria:

* A diagnosis of substance dependence (DSM-IV)
* Known allergy to study medication
* Currently taking warfarin or having anamnestic indicators of impaired haemostasis (profuse bleeding, except epistaxis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2001-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS)- Total | Baseline - 8 weeks - 16 weeks

SECONDARY OUTCOMES:
PANSS Subscales Negative, Positive, General Psychopathology | Weeks 0, 8, 16
GLOBAL ASSESSMENT OF FUNCTIONING- Split Version (S-GAF) | Weeks 0, 8, 16
  (S-GAF)Symptom Scale (S-GAF)Function Scale
WONCA-COOP FUNCTIONAL HEALTH ASSESSMENT CHARTS | Weeks 0, 8, 16
  5 scales
NIACIN SKIN FLUSH TEST | Weeks 0, 8, 16
  2 concentrations of niacin
THE UKU SIDE EFFECT RATING SCALE (USERS) | Weeks 0,4,8,12,16
  1. Sum of scores
  2. Patients with side effects
SERIOUS ADVERSE EVENTS | Weeks 0,4,8,12,16
CONCOMITANT ANTIPSYCHOTIC MEDICATION | Weeks 0,4,8,12,16
  Defined Daily Doses (ATC/WHO)
Kimura Recurring Recognition Figures Test | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Hopkins Verbal Learning Test. | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Continuous Performance Test | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Hopkins Verbal Learning Test | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Paced Auditory Serial Addition Test | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Stroop Test | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Digit Span | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
The Letter - Number Task | Weeks 0,16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Semantic and Category Fluency | Weeks 0, 16
  A sub-sample of patients. For logistic reasons, only some study sites could participate.
Body Mass Index | Weeks 0, 16
Blood pressure - systolic, diastolic | Weeks 0, 16
Heart rate | Weeks 0, 16
Albumin | Weeks 0, 16
  Serum
Urate | Weeks 0, 16
  Serum
Glucose | Weeks 0, 16
  Serum - fasting
Cholesterol | Weeks 0, 16
  Serum - fasting
Triglycerides | Weeks 0, 16
  Serum - fasting
Fatty acids in red blood cells | Weeks 0, 16
  The concentrations of long-chain (C14-18) and very long-chain (C20-24)fatty acids in erythrocytes were measured. Fasting condition.
  We selected DGLA, AA, EPA, DHA, total omega-3 Polyunsaturated Fatty Acids (PUFA), total omega-6 PUFA, PUFA and LCPUFA (long-chain PUFA) as outcome measures.
Alpha-tocopherol adjusted for [triglycerides]+[cholesterol]. | Weeks 0, 16
  Serum
Total antioxidant status | Weeks 0, 16
  Serum
Malondialdehyde | Weeks 0, 16
  Also called "TBARS". Serum
F2-isoprostane (8-epiPGF2-alpha) | Weeks 0, 16
  Serum
Cytosolic PLA2 group IV in red blood cells(ELISA method)
  Omitted from stastical analyses because of problems with the pre-analytic procedure (treatment the of blood)
Gene expression of mRNA for Phospholipase A2 (PLA2) groups IVa and VIa in monocytes. | Weeks 0, 16
  Whole blood
Mean Corpuscular Haemoglobin Concentration (MCHC) | Weeks 0, 16
  Whole blood
Mean Corpuscular Volume (MCV) | Weeks 0, 16
  Whole blood
C- Reactive Protein (CRP) | Weeks 0, 16
  Plasma
Haemoglobin | Weeks 0, 16
  Whole blood
Leukocytes | Weeks 0, 16
  Whole blood
Calcium | Weeks 0, 16
  Serum
Sodium | Weeks 0, 16
  Serum
Potassium | Weeks 0, 16
  Serum
Ferritin | Weeks 0,16
  Serum
Free thyroxin (T4) | Weeks 0, 16
  Serum
Thyroid Stimulating Hormone (TSH) | Weeks 0, 16
  Serum

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Bentsen, MD PhD, Study Director — Aker University Hospital (-2004), Diakonhjemmet Hospital (2004-); Odd Lingjærde, MD PhD, Study Chair — University Hospital, Aker
Locations (1):
- Aker University Hospital, Oslo, Norway